CLINICAL TRIAL: NCT05841901
Title: Evaluation of the Efficacy and Mechanism of Action of Huang-long Zhi-xiao Granule to Improve the Control Rate of Chronic Persistent of Asthma
Brief Title: Huang-long Zhi-xiao Granule Improves the Control Rate of Chronic Persistent of Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for Asthma
Record Dates: First submitted 2023-02-03; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Asthma Chronic
Keywords: Huang-long Zhi-xiao Granule; Chronic persistent of asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huang-long Zhi-xiao Granule (Experimental): Huang-long Zhi-xiao Granule, Honey ephedra 6g, shot dried 10g, earth dragon 10g, Ganoderma lucidum 20g, Qianhu 12g, perilla seed 10g, Zhejiang fritillary 9g, soaphorn thorn 9g, scorched mulberry white peel 20g, fried white nuts 10g, fructus nume 10g, licorice 6g.
  Interventions: Drug: Huang-long Zhi-xiao Granule
- Huang-long Zhi-xiao Granule placebo (Placebo Comparator): The Huang-long Zhi-xiao Granule placebo is prepared by adding 5% of the drug on the basis of dextrin and bitter agent, and its appearance, weight, color and smell are consistent with Chinese medicine granules.
  Interventions: Drug: Huang-long Zhi-xiao Granule placebo

INTERVENTIONS:
Drug: Huang-long Zhi-xiao Granule — The experimental group was given Huang-long Zhi-xiao Granule.1 dose per day, oral in 2 divided doses, 1 course every 4 weeks, for a total of 8 weeks of treatment.
  Arms: Huang-long Zhi-xiao Granule
Drug: Huang-long Zhi-xiao Granule placebo — The toncral group was given placebo Huang-long Zhi-xiao Granule.The course of treatment was the same as that of the experimental group.
  Arms: Huang-long Zhi-xiao Granule placebo

SUMMARY:
The goal of this observational study is to test the Evaluation of the efficacy and mechanism of action about Huang-long Zhi-xiao Granule to improve the control rate of Asthma chronic duration. The main questions it aims to answer are:

* [Relying on the top-level experimental design, scientifically evaluated the efficacy and safety of Huang-long Zhi-xiao Granule in patients with chronic asthma (hot asthma), and provided evidence support for the clinical application of Classical Prescriptions.]
* [Through the retained sample to test Asthma-related inflammatory indicators, immunoglobulins, T cell subsets, etc. To investigate the mechanism of action of Huang-long Zhi-xiao Granule in patients with chronic duration of asthma (hot asthma).]

DETAILED DESCRIPTION:
Bronchial asthma attacks are erratic and difficult to heal, which seriously affects the quality of life of patients, and their physical and mental health is also seriously affected by asthma.

This study will conduct clinical observations in patients with chronic persistence (hot wheezing) of bronchial asthma, scientifically evaluate the efficacy and safety of Huanglong Anti-Wheezing in patients with asthma chronic duration (hot wheezing), and provide evidence support for the clinical application of Huanglong Anti-Wheezing Formula.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for chronic persistent bronchial asthma
* It meets the TCM differentiation standards for wheezing and hot wheezing
* Asthma Control Test (ACT) questionnaire score<20 score
* The severity of disease is graded from mild to moderately persistent
* Patients who have not been treated with anti-asthmatic drugs for 2 weeks prior to dosing or who have been treated with ICS or ICS+LABA for 4 weeks or more prior to dosing and who have the same type and dose of the drug
* Age form 18-80 years old
* Have not participated in other clinical studies within 1 month prior to enrollment
* Voluntarily participate in the study and sign an informed consent form

Exclusion Criteria:

* Patients with special types of refractory asthma, critical asthma, occupational asthma, seasonal asthma, atypical asthma or tuberculosis, pulmonary interstitial fibrosis, thoracic malformation, chronic obstructive pulmonary disease, bronchiectasis, cystic pulmonary fibrosis, allergic bronchopulmonary aspergillosis, allergic granulomatous vasculitis, infectious, restrictive lung disease and other airflow obstructive pulmonary diseases
* Patients with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina, acute myocardial infarction, cardiac function grade 3 and above, stroke, cerebral hemorrhage, etc.)
* Glutamate aminotransferase (ALT), aspartate aminotransferase (AST) > 1.5 times the upper limit of normal value， blood creatinine (Cr) > upper limit of normal value
* Those who are allergic and allergic to the components of drugs in known test drugs
* Patients with bronchiectasis, tuberculosis, pulmonary embolism, or other serious respiratory conditions
* Combined with severe cognitive and psychiatric abnormalities
* Participants who are pregnant, lactating, and planning to become pregnant
* Those who are participating in other clinical trials within 1 month prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Asthma control tests（CAT） | Change from baseline CAT scores at week 4, 8, 21, 34，47 and 52.
  CAT will be used to evaluate quality of life. A total score of 0-40 will be given with a higher score indicating a worse condition.
Frequencies of acute attacks | Up to week 52.
  It will be assessed by frequencies of asthma-related hospitalizations.The patient's disease progression was recorded by recording the number of acute attacks at each time point, as well as the specific condition at the time of the attack.

SECONDARY OUTCOMES:
Asthma exacerbation severity and hospitalization rate | Week0(before treatment),week4、week8、week21、week34、week47and week52.
  Worsening lung function during asthma attacks is characterized by decreased expiratory flow, and the severity of the exacerbation can be graded by the patient's symptoms, lung function, and arterial blood gas analysis.According to the frequency of daytime and nighttime asthma attacks and pulmonary function test results, the patients were divided into 4 grades, namely: 1 intermittent attack; 2 mild persistent; 3 moderate persistent and 4 severe persistent.The severity of the asthma attack was assessed using a rating scale
Change in severity of chronic persistent disease | Week0(before treatment),week4、week8、week21、week34、week47and week52.
  Although the patient does not have an acute attack of asthma, there are still symptoms such as wheezing, cough, chest tightness and other symptoms with different frequency and degrees for a long time, which may be accompanied by decreased pulmonary ventilation function. The severity of chronic persistent asthma can be classified into four levels: intermittent, mildly persistent, moderately persistent, and severely persistent, according to the frequency of daytime and nighttime asthma symptoms and the results of pulmonary function tests.The severity of the asthma attack was assessed using a rating scale
The dose used by glucocorticoids | Week0(before treatment),week4、week8、week21、week34、week47 and week52.
  Corticosteroids are the drug of choice for long-term asthma treatment. The vast majority of patients with chronic persistent asthma are well controlled by inhaling low-dose corticosteroids (equivalent to 400 micrograms of budesonide per day).
Rapid-acting beta2 agonists use drugs and doses | Week0(before treatment),week8 and after follow-up（week52）
  Beta2 agonists are asthma drugs that stimulate beta2 receptors distributed on airway smooth muscle to produce bronchodilating effects. These drugs are bronchodilators and are the drugs of choice for acute asthma attacks (airway spasm), which can quickly improve symptoms such as dyspnea, cough, etc. If given by inhalation, salbutamol 100-200mcg or terbutaline 250-500mcg at a time and repeat every 20 minutes if necessary,
Score for clinical signs and symptoms | Week0(before treatment),week8 and after follow-up（week52）
  Formulate with reference to the "Guidelines for Clinical Research of New Chinese Medicines"Clinical scoring is weighted or assigned according to some of the main symptoms, signs, physiological parameters of patients, etc., so as to quantitatively evaluate the severity of the disease.The higher the score, the worse the state.
Pulmonary function | Week0(before treatment),week4、week8、week21、week34、week47and week52.
  Pulmonary function tests are an important part of the assessment of asthma and use objective indicators of lung function to monitor asthma.Routine pulmonary ventilation tests should be performed in all patients with clinically suspected asthma, and bronchodilator tests may be performed if ventilatory function suggests an obstructive change in ventilation. If the diastolic test is positive, the diagnosis of asthma can be established combined with clinical history, if the diastolic test is negative and FEV1 & GT. 70% predicted value, the conditional unit can do bronchial provocation test.
Exhaled nitric oxide | Week0(before treatment),week4、week8、week21、week34、week47and week52.
Asthma Control Questionnaire (ACQ) | Week0(before treatment),week8 and after follow-up（week52）
  The content of ACQ involves the following aspects: asthma-related, symptoms, the use of first-aid drugs, the impact on daily life and lung function test results.The higher the score, the worse the state.
Asthma Quality of Life Score (AQLQ) score | Week0(before treatment),week8 and after follow-up（week52）
  The asthma quality of life scale (5-point scale-RRB- consists of 35 items, including activity limitation (1-12) , asthma symptoms (13-20) , psychological status (22-26) , response to stimuli (27-31) , concern for one's own health (32-35) . On a 5-point scale, 1 is the worst and 5 is the best.
Sputum detection indicators | Week0(before treatment), week 8，after follow-up（week52）
  ①Induced sputum inflammatory phenotype: the inflammatory phenotype was classified into eosinophilic asthma, neutrophil asthma, paucigranulocytic asthma and mixed granulocytic asthma according to the detection of Eos in sputum②Eosinophil granulocyte cationic protein（EPC）③Inflammatory factors: IL-4, IL-5, Il-13, IL-25④Mucin MUC5AC.

CONTACTS AND LOCATIONS:
Overall Officials: Minghang Wang, MD, Principal Investigator — Henan University of Traditonal Chinese Medicine

IPD SHARING:
Plan to Share IPD: No